CLINICAL TRIAL: NCT05877014
Title: Unipolar Versus Bipolar Interlocking in Humeral Shaft Fractures in Adults
Acronym: UNILOCH
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MARTZ PHRCN 2021
Record Dates: First submitted 2023-05-17; First posted 2023-05-26 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Humeral Shaft Fracture
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Unipolar interlocking group (Experimental)
  Interventions: Other: questionnaires; Other: scanner
- Bipolar interlocking group (Active Comparator)
  Interventions: Other: questionnaires; Other: scanner

INTERVENTIONS:
Other: questionnaires — EQ-5D-5L and SF-12
Other: scanner — CT scan at M9 and then at M12 if the humerus is not consolidated at M6

SUMMARY:
Shaft fractures account for 20% of humeral fractures and 3% of all adult fractures in France, with an estimated incidence of 13 to 20/100,000 people. Men aged 21 to 30 years and women aged 60 to 80 years are particularly affected. Intramedullary nailing is among the standard treatments for humeral shaft fractures (when surgery is required). Once inserted, the nail is locked in order to limit stress on the fractured bone, as well as possible secondary rotational displacements or malunion. Bipolar interlocking (BI) is typically performed on both sides (proximal and distal) of the fracture site. This procedure is performed under radiological control, exposing the patient and care team to radiation (during the entire procedure). The objective of the treatment is to obtain consolidation of the fracture within 12 months, and to limit the occurrence of irreversible complications such as malunion or nonunion (2-10% at 12 months post-surgery). The "unipolar interlocking" (UI) technique has recently been introduced. In this technique, locking is performed only on the proximal side of the fracture site. By avoiding the distal approach, potential complications such as radial nerve damage, with the risk of irreversible paralysis (3.8-14.2% in studies of the BI technique in this indication) or the risk of infection on the distal side can be avoided. It also reduces operative time, and consequently the radiation received by patients and caregivers. However, the UI may be poorly positioned, resulting in malunion that requires revision surgery.

Despite the absence of recommendations due to the lack of existing data, several teams use the UI in routine care. In this context, a descriptive cohort of 121 patients operated on at the Dijon University Hospital5 showed similar rates of consolidation between the 2 techniques (93.8% for UI versus 95.2% for BI, p=0.64), functional scores, and complications, as well as a significant 29% decrease in operating time in the UI group (mean + SD: 63.1±21.3 min versus 88.0±30.1 min for VB, p<0.01). These encouraging results, although limited by the retrospective and observational nature of the data, justify a prospective randomized trial comparing these two techniques.

ELIGIBILITY:
Inclusion Criteria:

* Patient with written consent
* Patient ≥18 years of age with a diagnosis of humeral shaft fracture (all types in the AO classification) requiring surgical treatment with intramedullary nailing

Exclusion Criteria:

* Person not affiliated to national health insurance
* Patient unable to attend all study visits
* Patient with a pathologic fracture
* Patient with a post-traumatic brachial plexus injury at the time of inclusion
* Patient under court protection, guardianship or legal guardianship
* Pregnant, parturient or breastfeeding woman
* Patient admitted for revision surgery of a humerus fracture (insufficient healing or complication)
* Patient with an acute or chronic, unstable or poorly controlled disease that may interfere with the evaluation of the study objective, as determined by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2023-07-03 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with radiologically assessed bone healing at 12 months | Through study completion, an average of 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France

IPD SHARING:
Plan to Share IPD: No